CLINICAL TRIAL: NCT06819657
Title: Remote Ischemic Conditioning for Safety, Feasibility, and Preliminary Efficacy in Patients With Aneurysmal Subarachnoid Hemorrhage After Aneurysm Clipping: An Open-Label, Evaluator-Blinded Randomized Controlled Trial
Brief Title: Safety , Feasibility and Preliminary Efficacy of Remote Ischemic Conditioning in Patients With Aneurysmal Subarachnoid Hemorrhage After Aneurysm Clipping
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HX-B-2024033
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal; Cerebrovascular Disorders; Brain Diseases; Stroke; Cardiovascular Diseases; Vascular Diseases; Nervous System Diseases
MeSH Terms: conditions — Subarachnoid Hemorrhage; Cerebrovascular Disorders; Brain Diseases; Stroke; Cardiovascular Diseases; Vascular Diseases; Nervous System Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Other): Guideline-based therapy
  Interventions: Other: Guideline-based therapy
- RIC Group (Experimental): Guideline-based therapy + RIC (200 mmHg, bid, 7d)
  Interventions: Device: Remote Ischemic Conditioning Treatment Instrument; Other: Guideline-based therapy

INTERVENTIONS:
Device: Remote Ischemic Conditioning Treatment Instrument — Remote ischemic conditioning (RIC) was administered twice daily to the unilateral lower limb using a blood pressure cuff inflated to 200 mmHg for 7 consecutive days post-clipping
  Arms: RIC Group
Other: Guideline-based therapy — Guideline-based therapy

SUMMARY:
This study was designed to evaluate the safety and efficacy of remote ischemic conditioning (RIC) in patients with aneurysmal subarachnoid hemorrhage (aSAH) following surgical clipping.

Aneurysmal subarachnoid hemorrhage is a life-threatening condition that occurs when a cerebral aneurysm ruptures, causing bleeding into the subarachnoid space. Surgical clipping of the aneurysm is a standard procedure used to stop the bleeding and prevent re-rupture, thereby stabilizing the patient's condition.

Remote ischemic conditioning (RIC) is a non-invasive treatment that involves using a blood pressure cuff to induce brief, temporary cycles of ischemia and reperfusion in a limb. Research suggests that this process may confer systemic protective effects, potentially improving recovery from brain injury or surgery. Although RIC has shown potential to improve outcomes in patients with other neurological conditions, its effect on patients with aSAH who undergo surgical clipping remains unclear.

This study will evaluate whether RIC can reduce complications, improve neurological function, and enhance overall recovery in these patients. The findings will help determine whether RIC should be incorporated into the standard treatment regimen for aSAH.

ELIGIBILITY:
Inclusion Criteria:

1. Imaging examination confirmed aneurysmal subarachnoid hemorrhage.
2. Responsible aneurysms received craniotomy clipping within 24 hours.
3. 18≤ age ≤80 years old.
4. Informed consent of the participant or legally authorized representative

Exclusion Criteria:

1. Patients with other types of cerebral hemorrhage.
2. Prior neurological impairment (mRS Score >1) or mental illness may confuse neurological or functional assessment.
3. Severe comorbidities with a life expectancy of less than 90 days.
4. Refractory hypertension (systolic blood pressure 180>mmHg or diastolic blood pressure 110>mmHg).
5. RIC contraindications: severe soft tissue injury of lower limbs.
6. Simultaneously participate in another research program to study a different experimental therapy.
7. Any condition that the investigator believes may increase the patient's risk.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of mRS (0-2) | 90±7 days post-enrollment in the study
  Modified Rankin Scale, mRS; min:0, max:6; A smaller score indicates a better prognosis.
incidence rate of RIC adverse events | From enrollment to the end of RIC at 1 week
  RIC adverse events mainly include: limb pain, skin damage, deep vein thrombosis, transient hypertension, etc.

SECONDARY OUTCOMES:
mRS Score as ordinal variable | 7±1 days post-enrollment in the study
  Modified Rankin Scale, mRS; min:0, max:6; A smaller score indicates a better prognosis.
mRS Score as ordinal variable | 30±7 days post-enrollment in the study
  Modified Rankin Scale, mRS; min:0, max:6; A smaller score indicates a better prognosis.
incidence rate of aSAH complications | From enrollment to 90 days post-enrollment
  The complications of aneurysmal subarachnoid hemorrhage mainly include cerebral vasospasm, delayed cerebral ischemia, hydrocephalus, rebleeding, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xu L, Jin T, Niu H, Yin Y, Yan K, Guan H, Liu A. Remote ischemic conditioning for safety, feasibility and preliminary efficacy of patients with aneurysmal subarachnoid hemorrhage after aneurysm clipping, design, and protocol for an open-label, evaluator blinding randomized controlled trial. Front Neurol. 2025 Nov 20;16:1650773. doi: 10.3389/fneur.2025.1650773. eCollection 2025. PMID 41356238